CLINICAL TRIAL: NCT06629883
Title: Personalized Resistance Training with Peer Support for Women with PCOS Using a Smart Home Video Device: Feasibility Study Guided by Self-Determination Theory
Brief Title: Resistance Exercise and Peer Support with Bands/balls and Digital Support Among Women with Polycystic Ovary Syndrome
Acronym: REPS w/BANDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Pamela J. Wright, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00120540
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: polycystic ovary syndrome; motivation; resistance training; digital technology; proof of concept study; feasibility studies
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- REPS w/BANDS (Experimental): The intervention was delivered by certified personal trainers who connected with participants in their homes using SHVDs. Supervised training was individually delivered to participants in real time and incorporated low-cost, portable resistance equipment (i.e., resistance bands, stability ball). SDT-guided strategies (e.g., peer support, practice, encouragement, affirmations) were incorporated to help increase exercise motivation. Peer support was addressed by randomly assigning participants with a buddy. Personal trainers demonstrated proper exercise form and had participants practice each exercise. Participants were instructed on how to use an affirmation app on the SHVD and encouraged to use it at least weekly.
  Interventions: Behavioral: REPS w/BANDS

INTERVENTIONS:
Behavioral: REPS w/BANDS — This theory-informed, one-arm proof-of-concept study provided participants (n=10) with an SHVD, exercise equipment (exercise bands, stability ball), and 2 supervised RE sessions per week for 12 weeks via the SHVD's video feature and incorporated strategies from self-determination theory to meet the psychological needs of autonomy, competence, and relatedness. Participants were randomly paired with a buddy.

SUMMARY:
The purpose of this one arm pilot was to assess the feasibility and acceptability of REPS w/BANDS and evaluate for signals of improvement for depressive symptoms, anthropometrics, and muscular endurance. Participants completed a 12-week personalized in-home resistance exercise program that was delivered in real-time via a smart home video device along with a buddy system for peer support.

DETAILED DESCRIPTION:
Research findings reveal that women with polycystic ovary syndrome (PCOS) report low exercise motivation due to PCOS stigma-related stress and lack of social connection, thus inhibiting exercise in public and group settings. The purpose of this study was to implement and assess the feasibility and acceptability of an in-home personalized resistance exercise (RE) program delivered in real time by a smart home video device (SHVD) with peer support provided by a buddy system. This theory-informed, one-arm proof-of-concept study provided participants (n=10) with an SHVD, exercise equipment (exercise bands, stability ball), and 2 supervised RE sessions per week for 12 weeks via the SHVD's video feature and incorporated strategies from self-determination theory to meet the psychological needs of autonomy, competence, and relatedness. Participants were randomly paired with a buddy. Feasibility, acceptability, depressive symptoms, anthropometrics, and muscular endurance were measured using surveys, fitness testing, and interviews. Quantitative data were calculated using t-tests. Qualitative data were analyzed via thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* an age of 18 or older
* a confirmed PCOS diagnosis by a healthcare provider
* physical activity readiness as determined by the Physical Activity Readiness Questionnaire (PAR-Q)
* residence within driving distance of the main university campus.

Exclusion Criteria:

* cardiorespiratory disease (e.g., congestive heart failure)
* hypertension
* orthopedic injury (e.g., herniated disc)
* pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | At the end of 12 weeks
  Screened participants # / Enrolled participants #
Attendance | At the end of 12 weeks
  Session # attended / Session # prescribed
Retention | At the end of 12 weeks
  Participant # completing 2nd assessment / Participant # completing baseline assessment
Acceptability Interviews | At the end of 12 weeks
  Acceptability was measured via content analysis of participant interviews
Acceptability Likert Scales | At the end of 12 weeks
  Questions of about satisfaction with REPS w/BANDS were scored on a scale of 0-4, with O indicating poor and 4 indicating excellent.

SECONDARY OUTCOMES:
Depressive Symptoms | From baseline and at the end of 12 weeks
  he Personal Health Questionnaire (PHQ-8) was used to assess prevalence and severity of depressive symptoms occurring within the past two weeks. The score is the sum of the 8 items. 0-4 = minimal or no depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-24 = severe depression
Bodyweight | At baseline and at the end of 12 weeks
  Participants self-reported body weight in pounds during the fitness assessments.
Height | At baseline and at the end of 12 weeks
  Participants self-reported height in feet and inches during the fitness assessments.
Waist Circumference | At baseline and at the end of 12 weeks
  Participants were guided to measure waist circumference in inches during the fitness assessments.
Squat Test | At baseline and at the end of 12 weeks
  Lower body muscular endurance was measured using the squat test. The score was the number of squats performed with proper form.
Modified Push Up Test | At baseline and at the end of 12 weeks
  Upper body muscular endurance was measured with this test. The score was the number of correctly performed push-up in one minute.
Curl Up Test | At baseline and at the end of 12 weeks
  This test was used to measure muscular endurance of the core. The score was the number of curl up properly performed to a cadence of 40bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Wright, PhD, MS, MEd, Principal Investigator — University of South Carolina
Locations (1):
- Clinical Exercise Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD was not shared to maintain participant confidentiality. Participants were assigned a unique identifier. All data was secured on university research servers that have multiple fire walls and are password protected. Source documents are stored in locked filing cabinets in a locked office in the College of Nursing. Source data have the participant identifier only. Findings will be reported in aggregate form.

REFERENCES:
- [Background] Wright PJ, Corbett CF, Pinto BM, Dawson RM, Wirth M. Resistance Training as Therapeutic Management in Women with PCOS: What is the Evidence? Int J Exerc Sci. 2021 Aug 1;14(3):840-854. doi: 10.70252/NEEX8658. eCollection 2021. PMID 34567361
- [Background] Behboodi Moghadam Z, Fereidooni B, Saffari M, Montazeri A. Measures of health-related quality of life in PCOS women: a systematic review. Int J Womens Health. 2018 Aug 1;10:397-408. doi: 10.2147/IJWH.S165794. eCollection 2018. PMID 30123008
- [Background] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Background] Azziz R. Epidemiology and pathogenesis of the polycystic ovary syndrome in adults. 2020. http://www.uptodate.com/contents/epidemiology-and-pathogenesis-of-the-polycysticovary-syndrome/